CLINICAL TRIAL: NCT06981390
Title: Ticagrelor-Based Dual Antiplatelet Therapy in Coronary Artery Bypass Grafting: A Randomized Clinical Trial on Graft Patency
Brief Title: Ticagrelor-Based Dual Antiplatelet Therapy Duration in CABG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kexiang Liu, MD (Other)
Responsible Party: Sponsor-Investigator, Kexiang Liu, MD, Principal Investigator, Second Hospital of Jilin University
Organization: Second Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JDEYXWK2025146
Record Dates: First submitted 2025-05-02; First posted 2025-05-20 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Grafting; Saphenous Vein; Dual Antiplatelet Therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Aspirin; 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3-Month DAPT Group (Active Comparator): Ticagrelor (90 mg BID) + Aspirin (100 mg QD) for 3 months, followed by aspirin monotherapy
  Interventions: Drug: Ticagrelor + Aspirin for 3 Months (followed by aspirin monotherapy)
- 6-Month DAPT Group (Active Comparator): Ticagrelor (90 mg BID) + Aspirin (100 mg QD) for 6 months, followed by aspirin monotherapy
  Interventions: Drug: Ticagrelor + Aspirin for 6 Months (followed by aspirin monotherapy)
- 12-Month DAPT Group (Experimental): Ticagrelor (90 mg BID) + Aspirin (100 mg QD) for 12 months, followed by aspirin monotherapy
  Interventions: Drug: Ticagrelor + Aspirin for 12 Months (followed by aspirin monotherapy)

INTERVENTIONS:
Drug: Ticagrelor + Aspirin for 3 Months (followed by aspirin monotherapy) — Ticagrelor (90 mg BID) + Aspirin (100 mg QD) for 3 months, followed by aspirin monotherapy
  Other Names: 3-Month DAPT
  Arms: 3-Month DAPT Group
Drug: Ticagrelor + Aspirin for 6 Months (followed by aspirin monotherapy) — Ticagrelor (90 mg BID) + Aspirin (100 mg QD) for 6 months, followed by aspirin monotherapy
  Other Names: 6-Month DAPT
  Arms: 6-Month DAPT Group
Drug: Ticagrelor + Aspirin for 12 Months (followed by aspirin monotherapy) — Ticagrelor (90 mg BID) + Aspirin (100 mg QD) for 12 months, followed by aspirin monotherapy
  Other Names: 12-Month DAPT
  Arms: 12-Month DAPT Group

SUMMARY:
This randomized controlled trial aims to evaluate the impact of different durations of Ticagrelor-based dual antiplatelet therapy (DAPT) on saphenous vein graft (SVG) patency in patients undergoing coronary artery bypass grafting (CABG). A total of 300 patients will be randomly assigned to receive Ticagrelor (90 mg BID) + Aspirin (100 mg QD) for 3 months, 6 months, or 12 months, followed by aspirin monotherapy.The primary outcome is 1-year graft patency, assessed via coronary CT angiography. Secondary outcomes include bleeding events (BARC classification), major adverse cardiovascular and cerebrovascular events (MACCE), and all-cause mortality. The study aims to determine the optimal DAPT duration to balance graft patency benefits and bleeding risks, ultimately guiding postoperative antiplatelet strategies for CABG patients.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is a widely used revascularization strategy for patients with complex coronary artery disease. However, the long-term patency of saphenous vein grafts (SVGs) remains a significant clinical concern, with graft occlusion being a major contributor to recurrent ischemic events. Dual antiplatelet therapy (DAPT), consisting of Ticagrelor and Aspirin, is commonly used to prevent thrombosis and improve graft patency, yet the optimal duration of DAPT post-CABG remains unclear. This randomized, double-blind, controlled trial aims to assess the effects of different DAPT durations on SVG patency and clinical outcomes in CABG patients. A total of 300 patients undergoing isolated CABG with at least one SVG will be enrolled and randomly assigned (1:1:1) to receive Ticagrelor (90 mg BID) + Aspirin (100 mg QD) for 3 months, 6 months, or 12 months, followed by aspirin monotherapy. The primary outcome of the study is SVG patency at 12 months, assessed via coronary CT angiography, defined as FitzGibbon Grade A (≤50% stenosis). Secondary outcomes include bleeding events , major adverse cardiovascular and cerebrovascular events (MACCE), and all-cause mortality. Patients will be followed at 3, 6, and 12 months postoperatively, undergoing clinical assessments, laboratory tests, and imaging evaluations to monitor graft patency, bleeding complications, and cardiovascular and cerebrovascular events. The study will provide critical data to determine the optimal duration of DAPT to maximize graft patency while minimizing bleeding risks, ultimately guiding personalized antiplatelet strategies in CABG patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-80 of age.
2. Patients undergo planned CABG for the first time with ≥1 SVGs
3. Patients with written informed consent.

Exclusion Criteria:

1. Patients undergoing concomitant valve surgery (excluding aortic bioprosthesis), aortic surgery, or rhythm surgery during the same session.
2. Patients undergoing emergency CABG.
3. Patients with single-vessel coronary artery disease.
4. Patients with cardiogenic shock or hemodynamic instability.
5. Patients with sick sinus syndrome, second- or third-degree atrioventricular block.
6. Patients with contraindications for coronary computed tomography angiography (CCTA) or coronary angiography, including contrast media allergy.
7. Patients requiring antiplatelet therapy other than aspirin or ticagrelor (e.g., clopidogrel, prasugrel) and unable to discontinue such medication after CABG, based on physician or investigator judgment.
8. Patients on oral anticoagulants before CABG who must continue anticoagulation therapy postoperatively.
9. Patients with contraindications for ticagrelor or aspirin, including:

   9.1Bleeding diathesis within the past 3 months. 9.2Severe gastrointestinal bleeding within the past year. 9.3Peptic ulcer (even without bleeding) within the past 3 years. 9.4History of intracranial hemorrhage, aspirin allergy, or severe aspirin-induced gastrointestinal reaction.
10. Patients with a drug-eluting stent (DES) in a coronary or cerebral artery within 6 months before CABG, or a bare-metal stent (BMS) within 1 month before CABG.
11. Patients with thrombocytopenia (<100 x 10⁹/L) before CABG.
12. Patients with severe renal dysfunction requiring dialysis or active liver disease, including unexplained persistent transaminase elevation or transaminase levels >3× the upper normal limit.
13. Patients using strong CYP3A4 inhibitors.
14. Patients requiring methotrexate and ibuprofen therapy.
15. Patients with active malignant tumors with an increased risk of bleeding, as determined by the investigator.
16. Pregnant or breastfeeding women, and those who have given birth within the past 90 days.
17. Premenopausal women not using adequate contraception. Adequate contraception requires at least two reliable methods, including one barrier method.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Saphenous Vein Graft (SVG) Patency at 12 Months | 12 months post-CABG
  SVG patency will be assessed using coronary CT angiography, defined as FitzGibbon Grade A (≤50% stenosis). The patency rates will be compared among the three groups receiving Ticagrelor-based DAPT for different durations (3 months, 6 months, or 12 months).

SECONDARY OUTCOMES:
Bleeding Events | Up to 12 months post-CABG
  Bleeding events as defined by the BARC classification ≥ 2 at 1 year after CABG.
MACCE episodes | Within 1-year after CABG
  MACCE episodes within 1-year after CABG (composite of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke or revascularization), as defined by the American College of Cardiology and American Heart Association and judged by an independent Clinical Endpoint Committee blinded to treatment allocation
All-Cause Mortality | Up to 12 months post-CABG
  Death from any cause occurring during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: kexiang liu, Study Director — Second Hospital of Jilin University
Locations (1):
- the Second Hospital of Jilin University, Changchun, Jilin, China